CLINICAL TRIAL: NCT04982549
Title: A Prospective Study to Evaluate the Safety of Concurrent Durvalumab (MEDI4736) With Chemoradiation Therapy（CRT）Followed by Durvalumab for Chinese Unresectable Stage III Non Small Cell Lung Cancer（NSCLC）
Brief Title: A Study to Evaluate the Safety of Concurrent Durvalumab With CRT Followed by Durvalumab for Chinese Unresectable Stage III NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4191L00116
Record Dates: First submitted 2021-05-07; First posted 2021-07-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Unresectable Stage III NSCLC
MeSH Terms: interventions — durvalumab; CP protocol; Pemetrexed; Cisplatin; Carboplatin; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + platinum-based chemotherapy and radiation (Experimental): All patients will receive 1 of the following platinum-based standard of care chemotherapy options, based on Investigator discretion, in addition to radiation therapy:
  cisplatin/etoposide carboplatin/paclitaxel pemetrexed/cisplatin pemetrexed/carboplatin At the completion of standard of care chemoradiation therapy (SoC CRT), patients with complete response, partial response or stable disease will continue to receive durvalumab as consolidation treatment.
  Interventions: Drug: Durvalumab; Drug: Carboplatin/ Paclitaxel; Drug: Pemetrexed/ Cisplatin; Drug: Pemetrexed/ Carboplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (intravenous infusion)
  Other Names: MEDI4736
Drug: Carboplatin/ Paclitaxel — Carboplatin /Paclitaxel, as per standard of care
Drug: Pemetrexed/ Cisplatin — Pemetrexed / Cisplatin, as per standard of care
Drug: Pemetrexed/ Carboplatin — Pemetrexed / Carboplatin , as per standard of care
Radiation: Radiation — 5 fractions/ week for ~6 weeks (±3 days) (Total 60 Gy)

SUMMARY:
This is a prospective, multi-center, single arm study assessing the efficacy and safety of durvalumab given concurrently with platinum-based CRT (durvalumab + SoC CRT) in patients with locally advanced, unresectable NSCLC (Stage III).

DETAILED DESCRIPTION:
Approximately 35 patients with locally advanced, unresectable NSCLC (Stage III) who are eligible to receive platinum-based CRT will be enrolled in and receive durvalumab + SoC CRT. Patients with CR, partial response (PR), or stable disease (SD）based on Investigator assessment at the 16-week tumor evaluation following completion of SoC CRT will continue to receive durvalumab as consolidation treatment. Patients with RECIST 1.1-defined radiological progressive disease (PD) will proceed to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically-documented NSCLC
* Locally advanced, unresectable (Stage III) NSCLC
* World Health Organization (WHO) performance status 0-1
* At least one measurable lesion, not previously irradiated
* Must have a life expectancy of at least 12 weeks at randomization
* Adequate lung function: Pre- or post-bronchodilator forced expiratory volume 1 of 1.0 L or >40% predicted value and DLCO >30% predicted value
* Must provide an archived tumor tissue block(or at least 15 newly cut unstained slides)≤3 years old; if archived sample unavailable then must provide a recent(≤3 months) tumor biopsy.

Exclusion Criteria:

* Mixed small-cell and NSCLC histology
* Receipt of prior or current cancer treatment, including but not limited to, radiation therapy, investigational agents, chemotherapy, Durvalumab and mAbs.
* Prior exposure to immune-mediated therapy, including but not limited to, other anti- CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies.
* Patients whose radiation treatment plans are likely to encompass a volume of whole lung receiving ≥20 Gy in total (V20) of more than 35% of lung volume
* Planned radiation cardiac dose V50>25%
* Any medical contraindication of platinum-based doublet chemotherapy as listed in the local labelling or known allergy/hypersensitivity to investigational product and/or its excipients
* History of the following: allogeneic organ transplantation, active or prior autoimmune or inflammatory disorders, another primary malignancy, leptomeningeal carcinomatosis, active primary immunodeficiency
* Uncontrolled intercurrent illness or active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Grade ≥3 immune-mediated Adverse event | From the date of first dose until disease progression,assessed up to 4 years
  Grade ≥3 immune-mediated Adverse event

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first dose until the date of objective disease progression or death,assessed up to 4 years
  Progression-free survival
Overall Survival (OS) | From the date of first dose until death due to any cause,assessed up to 4 years
  Overall Survival
Objective response rate(ORR) | From the date of first dose until the date of objective disease progression or death,assessed up to 4 years
  Objective response rate
Duration of response(DOR) | From the date of first documented response (RECIST 1.1.) until the first date of documented progression or death in the absence of disease progression,assessed up to 4 years
  Duration of response
Disease control rate(DCR) | From the date of first dose until 24 weeks.
  Disease control rate
Time to death or distant metastasis(TTDM) | From the date of first dose to until the first date of distant metastasis or death in the absence of distant metastasis,assessed up to 4 years
  Time to death or distant metastasis

OTHER OUTCOMES:
Adverse events | From the date of enrollment until disease progression,assessed up to 4 years
  Adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality